CLINICAL TRIAL: NCT02392806
Title: Comparative Effectiveness Study of Bubble CPAP Devices in the NICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marya Strand, MD (Other)
Responsible Party: Sponsor-Investigator, Marya Strand, MD, Associate Professor, Pediatrics, St. Louis University
Organization: St. Louis University (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SLU Protocol # 24949
Record Dates: First submitted 2015-02-27; First posted 2015-03-19 (Estimated); Results first posted 2017-12-26 (Actual); Last update posted 2018-03-09 (Actual); Status verified 2018-02

CONDITIONS: Respiratory Distress Syndrome
Keywords: Continuous positive airway pressure; CPAP; Bubble CPAP; Extubation failure; Preterm infant
MeSH Terms: conditions — Respiratory Distress Syndrome; Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BabiPlus, Respiralogics (Active Comparator): Infants randomized to the BabiPlus device will be extubated to BabiPlus Bubble CPAP device and after 72 hours, if the infant has remained extubated, will be crossed-over to the B&B Bubbler device for 24 hours
  Interventions: Device: Bubble CPAP- BabiPlus, Respiralogics
- B&B Bubbler, B&B medical Technologies (Active Comparator): Infants randomized to the B&B Bubbler device will be extubated to B&B Bubbler Bubble CPAP device and after 72 hours, if the infant has remained extubated, will be crossed-over to the BabiPlus device for 24 hours
  Interventions: Device: Bubble CPAP- B&B Bubbler, B&B Medical devices

INTERVENTIONS:
Device: Bubble CPAP- BabiPlus, Respiralogics — Infant will be randomized to BabiPlus Bubbler at time of extubation
  Other Names: Bubble Continuous Positive Airway Pressure (BCPAP)
  Arms: BabiPlus, Respiralogics
Device: Bubble CPAP- B&B Bubbler, B&B Medical devices — Infant will be randomized to B&B Bubbler at time of extubation
  Arms: B&B Bubbler, B&B medical Technologies

SUMMARY:
Multiple different devices are available to provide Bubble CPAP to preterm and newborn infants. The most significant difference between these devices is the size of the bubble produced by the exhalation limb. This study will determine if one Bubble CPAP device (BabiPlus vs B&B) is more effective in improving oxygenation and decreasing extubation failure in the extremely low birthweight population.

DETAILED DESCRIPTION:
Primary outcome: Bubble CPAP failure (re-intubation or use of non-invasive positive pressure ventilation) within 72 hours following extubation Secondary outcome: Number of infants that reach 21% inspired oxygen during initial study period Secondary outcome: Apnea/bradycardia events in the initial study period Secondary outcome: Mean oxygen requirement following initial study period

Population: Infants born at <=1250 grams birth weight but >= 500 grams birth weight

Randomization: Equal allocation stratified by gestational age (<27 weeks, >=27 weeks)

Study diagram:

72h 24h X---------->X1----------->Y2 Y---------->Y1----------->X2 Infants will be randomly assigned to treatment X (BabiPlus, control group) or treatment Y (B&B Bubbler, intervention group). The primary outcome is bubble CPAP failure during the first 72 hours following extubation, measured at time point 1 in the diagram. Bubble CPAP failure is defined as requiring re-intubation or non-invasive positive pressure ventilation (NIPPV), requiring FiO2 of >60% for one hour or a pCO2 measurement of >65 mm Hg. For those infants that remain on CPAP during the initial study period, the number that reach 21% inspired oxygen for >12 consecutive hours will be compared between groups. This difference will also be analyzed using a Chi square test.

Those infants that remain on CPAP following the 72 hour initial study period (e.g., did not meet primary outcome criteria) will be crossed over to the opposite treatment arm for at least 24 hours. The minimum oxygen requirement required to keep the saturations in the ordered range, per standard NICU guidelines, will be recorded and compared between time points 1 and 2.

This study design is complex due to the nature of the disease of these patients. Each day every infant's premature pulmonary disease is evolving. There is no way to control for this.

ELIGIBILITY:
Inclusion Criteria:

1. Infant delivered at >=500 grams and <=1250 grams birth weight.
2. Infant requires intubation for mechanical ventilation within the first 48 hours following delivery.
3. Infant has received exogenous surfactant during mechanical ventilation.

Exclusion Criteria:

1. Decision by attending physician to redirect to comfort care
2. Congenital condition that precludes the use of CPAP (choanal atresia, diaphragmatic hernia, etc.)
3. Birth weight >1250 grams or <500 grams.
4. Non-English speaking parents. -

Ages: 1 Day to 100 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2015-01; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Noah H Hillman, M.D., Principal Investigator — Associate Director, Pediatrics
Locations (1):
- Cardinal Glennon Children's Hospital, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Bubble CPAP- BabiPlus, Respiralogics: Infants randomized to the BabiPlus device will be extubated to BabiPlus Bubble CPAP device and after 72 hours, if the infant has remained extubated, will be crossed-over to the B&B Bubbler device
  Bubble CPAP- BabiPlus, Respiralogics: Infant will be randomized to BabiPlus verses B&B Bubbler at time of extubation
- Bubble CPAP - B&B Bubbler, B&B Medical Technologies: Infants randomized to the B&B Bubbler device will be extubated to B&B Bubbler Bubble CPAP device and after 72 hours, if the infant has remained extubated, will be crossed-over to the BabiPlus device
  Bubble CPAP- B&B Bubbler, B&B Medical devices: Infant will be randomized to BabiPlus verses B&B Bubbler at time of extubation
Period: Overall Study
Arm/Group | Bubble CPAP- BabiPlus, Respiralogics | Bubble CPAP - B&B Bubbler, B&B Medical Technologies
Started | 22 | 21
Completed | 22 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bubble CPAP- BabiPlus, Respiralogics | Bubble CPAP - B&B Bubbler, B&B Medical Technologies | Total
Number analyzed (Participants) | 22 | 21 | 43
Age, Continuous [Mean (Standard Deviation); unit: Weeks Gestational Age] | 26.0 (2.0) | 25.4 (1.4) | 25.7 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 13 | 12 | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Extubation Failure
Description: Bubble CPAP failure (re-intubation or use of non-invasive positive pressure ventilation) within 72 hours following extubation
Time Frame: Within 72 hours of extubation
Measure: Count of Participants; unit: Participants
Arm/Group | Bubble CPAP- BabiPlus, Respiralogics | Bubble CPAP - B&B Bubbler, B&B Medical Technologies
Number analyzed (Participants) | 22 | 21
Participants | 9 | 7
Statistical Analysis 1: Comparison: Bubble CPAP- BabiPlus, Respiralogics vs Bubble CPAP - B&B Bubbler, B&B Medical Technologies; Test type: Superiority; p > 0.05, t-test, 2 sided

2. Secondary Outcome: Oxygenation - Oxygen Saturation Via Pulse Oximetry Recorded Hourly
Description: Number of infants that reach 21% inspired oxygen during initial study period of 72 hours plus the crossover period of 24 hours
Time Frame: 96 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Bubble CPAP- BabiPlus, Respiralogics | Bubble CPAP - B&B Bubbler, B&B Medical Technologies
Number analyzed (Participants) | 22 | 21
Participants | 5 | 5

ADVERSE EVENTS:
Arm/Group | Bubble CPAP- BabiPlus, Respiralogics | Bubble CPAP - B&B Bubbler, B&B Medical Technologies
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/21
Other Adverse Events (participants affected / at risk) | 0/22 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes